CLINICAL TRIAL: NCT00136136
Title: Validation of BIS-monitor in 3 Groups of Newborn Children
Brief Title: Validation of Bispectral Index (BIS)-Monitor in 3 Groups of Newborn Children
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2003/139
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal healthy term newborn: Normal healthy term newborns
  Interventions: Procedure: Registration of the bispectral index and spectral edge frequency
- Ill term newly born without brain damage: Ill term newly borns without brain damage
  Interventions: Procedure: Registration of the bispectral index and spectral edge frequency
- Preterm newly born without brain damage: Preterm newly borns without brain damage
  Interventions: Procedure: Registration of the bispectral index and spectral edge frequency

INTERVENTIONS:
Procedure: Registration of the bispectral index and spectral edge frequency — Registration of the bispectral index and spectral edge frequency

SUMMARY:
This study will evaluate the registration of the bispectral index and spectral edge frequency in relation to the behavioural state.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: normal healthy term newborns
* Group 2: Ill term newborns without brain damage
* Group 3: Preterm newborns without brain damage

Exclusion Criteria:

* Abnormal brain ultrasound
* Abnormal neurological examination
* Major congenital abnormalities
* Use of analgesics, sedatives, antiepileptic drugs or curarisation

Min Age: 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newborn children
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2003-08-01 (Actual); Primary Completion 2004-12-31 (Actual); Study Completion 2004-12-31 (Actual)

PRIMARY OUTCOMES:
Validation of the Bispectral Index(BIS)-Monitor | Short after birth of the newborn
  Validation of the Bispectral Index(BIS)-Monitor by registration of the bispectral index and spectral edge frequency in relation to behavioural state

CONTACTS AND LOCATIONS:
Overall Officials: Claudine De Praeter, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be